CLINICAL TRIAL: NCT06917326
Title: Clinical Pilot Study to Assess Safety and Performance of Neola®, a Novel Lung Monitoring Device for Neonates
Brief Title: Study to Assess Safety and Performance of Neola®, a Novel Lung Monitoring Device for Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neola Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PLN-0654; CIV-24-05-047374 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2025-03-14; First posted 2025-04-08 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: RDS of Prematurity; Preterm Birth; Lung Diseases
Keywords: GASMAS; Spectroscopy; Gas absorption spectroscopy
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Premature Birth; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Device: Monitoring

INTERVENTIONS:
Device: Monitoring — Lung monitoring with the Neola device

SUMMARY:
Clinical pilot study to assess safety and performance of Neola®, a novel lung monitoring device for neonates

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate that the device is safe and performs as intended under anticipated use conditions.

The performance of Neola will be evaluated in terms of ability to continuously measure and display the relative lung volume and absolute oxygen gas concentration on neonates. The results of this clinical investigation will provide further information for the design of a subsequent full-scale clinical investigation.

ELIGIBILITY:
Inclusion criteria:

* Preterm or term born neonates with gestational age between 28 and 40 weeks
* Post-natal age between 1 and 14 days
* Weight between 1000 g and 3000 g
* Signed informed consent prior to any study related procedures by the legal representatives of the patient
* Legal representatives are 18 years or older
* Legal representatives can absorb and understand the content of the informed consent form

Exclusion criteria:

* Known cardiopulmonary congenital anomalies
* Patients with trisomies or other chromosomal abnormality
* Patients not expected to survive
* Non-intact skin or other skin conditions (such as skin lesions) that do not allow the use of skin adhesives. (e.g., Bullous impetigo, Staphylococcal scalded skin syndrome, localized lesions of herpes simplex virus)
* Thorax curvature does not allow placement of the probe sets without air between the surface of the probes and the skin.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The number of serious and non-serious adverse events occurring during the trial | 2 days
  The primary objective of the study is to evaluate safety with regards to adverse events (AE) and in particular device related adverse events.
  Outcome measure: The number of serious and non-serious adverse events occurring during the trial.
The number of device related events including skin reactions | 2 days
  The primary objective of the study is to evaluate safety with regards to adverse events (AE) and in particular device related adverse events. Outcome measure: The number of device related events including skin reactions.

SECONDARY OUTCOMES:
The device's ability to continuously measure and present the clinical parameters while the neonates are in a resting state/sleeping | 2 hours
  This exploratory endpoint will be presented as the percentage of the total resting/sleeping time that the device is able to measure the clinical parameters relative lung volume and absolute oxygen concentration.
The device's ability to continuously measure and present the clinical parameters during normal handling of the neonates | 2 hours
  This exploratory endpoint will be presented as the percentage of the total handling time that the device is able to measure the clinical parameters relative lung volume and absolute oxygen concentration.
The adhesive performance of the probes in terms of ability to be repositioned and stay attached | 2 hours
  The adhesive performance of the probes in terms of ability to be repositioned and stay attached. This exploratory endpoint will be evaluated the percentage of probe adhesives that were able to stay attached for the duration of the measurement session.

OTHER OUTCOMES:
The gas absorption signals and noise at five different pre-determined locations of emitter and detector probe positions for the left and right side of the body | 2 hours
  The gas absorption is measured as %m, which is the gas concentration in % (partial pressure / total pressure) multiplied by absorption path length in meter (m). The signal to noise is measured as a ratio without any unit.
Influence of ambient light on the gas absorption signals | 2 hours
  This will be evaluated as how much ambient light contributes to the gas absorption signal, measured in the units %m. This will be evaluated by comparing gas absorption signals when ambient light is blocked versus not blocked.
  The gas absorption is measured as %m, which is the gas concentration in % (partial pressure / total pressure) multiplied by absorption path length in meter (m).
Influence of emitted light scattered out in the surrounding room that is detected by the detector probe | 2 hours
  This will be evaluated by assessing how much scattered light contributes to the gas absorption signal which is measured in the units %m. This will be evaluated by comparing gas absorption signals when scattered light is blocked versus not blocked.
  The gas absorption is measured as %m, which is the gas concentration in % (partial pressure / total pressure) multiplied by absorption path length in meter (m).

CONTACTS AND LOCATIONS:
Overall Officials: Gustaf Lernfelt, Principal Investigator — Sodra Alvsborgs Hospital
Locations (1):
- Södra Älvsborgs Sjukhus, Borås, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No